CLINICAL TRIAL: NCT03876925
Title: A Single Arm, Open-label,Phase Ib Study of CT053PTSA in Preciously Treated Patients With Advanced and Metastatic Renal Cell Cancer
Brief Title: A Single Arm, Open-label,Phase Ib Study of CT053PTSA in Preciously Treated Patients With Advanced and Metastatic RCC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The effect of CT053PTSA in preciously treated patients with advanced and metastatic RCC is not as good as pre-expected
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DCT053-17-001
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Renal Cell Cancer Metastatic
Keywords: RCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT053PTSA (Experimental): 60-100mg
  Interventions: Drug: CT053PTSA

INTERVENTIONS:
Drug: CT053PTSA — Patients will received oral CT053PTSA once daily until disease progression or intolerable toxicity or subject's withdrawal from treatment ,each cycle is defined as 28 days
  Other Names: Ningetinib

SUMMARY:
This is a phase Ib,single arm,open label study evaluating the safety and efficacy of CT053PTSA in patients with advanced and metastatic renal cell cancer who have progressed from previous treatment

DETAILED DESCRIPTION:
This study is being carried out in two parts,part 1 and part 2. Part 1: This is the dose-escalation part. The primary purpose of the part 1 portion is to determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD), and recommend the appropriate doses of CT053PTSA for further study Part 2: This is the expansion part.The part 2 portion of this study will continue to evaluate the safety and efficacy of CT053PTSA at the appropriate dose recommended in Part 1,in patients with advanced and metastatic RCC

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell cancer.Patients must be diagnosed with advanced or metastatic disease,disease progressed to previous treatment .
* Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Toxicity recovered to NCI CTCAE v.4.03 Grade ≤1 from previous treatments (except alopecia)
* ECOG performance status (PS) 0 or 1
* Life expectancy of ≥ 12 weeks
* Adequate organ function
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Chemotherapy,radiotherapy,immunotherapy and targeted therapy less than 4 months prior to administration.
* Symptomatic, untreated or unstable central nervous system metastases
* Uncontrolled hypertension that require anti-hypertensive agents to control, or systolic blood pressure (BP) >140mmHg or diastolic BP >90 mmHg before the first administration (BP is the mean blood pressure of two measures that 1 hours interval or above)
* Doppler ultrasound evaluation：Left ventricular ejection fraction < 50%
* Significantly clinical arrhythmia or symptomatic bradycardia, or male with QTCF > 450 ms or female with QTCF > 470 ms, or patients with a history of torsion or congenital QT prolonged syndrome long QT syndrome
* Certain factors that would preclude adequate absorption of CT053PTSA and gefitinib (eg. unable to swallow, chronic diarrhea, intestinal obstruction)
* Patients with evidence of bleeding tendency, including the following cases: gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above; or melena or hematemesis within 2 months; or visceral bleeding that may occur considered by investigator
* History of organ transplantation
* Any disease of the following bellowed within 12 months prior to administration: Myocardial infarction, severe angina, or unstable angina, coronary or peripheral artery bypass graft, congestive heart failure
* Pulmonary embolism or cerebrovascular events (including transient ischemic attack)within 6 months prior to administration
* Infection of HIV
* Patients with infection of HBV or HCV. Patients with positive of HBsAg or HBcAb,and HBV-DNA can be measured (>500IU/ml). Patients with positive of anti-HCV,and HCV-RNA can be measured by PCR.
* Other malignancies within 5 years prior to enrollment, with the exception of carcinoma in situ of the cervix, basal or squamous cell skin cancer
* Pregnant or lactating woman
* Any other reason the investigator considers the patient is not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Part 1(dose-escalation part):Maximum Tolerated Dose (MTD) | Cycle 1 Day 1 to Cycle 1 Day 28
  The maximum tolerated dose (MTD) of the CT053PTSA will be determined according to incidence of dose-limiting toxicity (DLT) assessed by NCI CTCAEv4.03
Part 2 (expansion part):Overall Response Rate | up to approximately 24 months
  Overall response rate (ORR),defined as a partial response (PR) or complete response (CR) occurring at any point post-treatment according to Response Evaluation Criteria in Solid Tumors as assessed by RECIST1.1

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) as a measure of safety and tolerability | up to approximately 24 months
  Safety and tolerability will be assessed through AEs, via monitoring changes in physical examination, clinical laboratory parameters, vital signs and ECGs
Disease Control Rate (DCR) | up to approximately 24 months
  DCR, proportion of patients with best overall response of CR, PR or SD
Progression-free Survival (PFS) | up to approximately 24 months
  PFS, defined as time from date of treatment to disease progression or death due to any cause
Duration of Response (DOR) | up to approximately 24 months
  DOR, defined as time from the first documented CR or PR to first documented progression or death due to any cause
Overall Survival (OS) | up to approximately 24 months
  OS, defined as time from date of treatment to death due to any cause
Maximum observed plasma concentration (Cmax) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile
Time of maximum observed plasma concentration (Tmax) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile
Area under the plasma concentration time curve (AUC) | Cycle 1 Day1 and Day 28
  to assess the pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Guo Jun, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No